CLINICAL TRIAL: NCT03845413
Title: Tobacco Control Network Among Women in Parana, Brazil - II
Brief Title: Gender-Relevant Tobacco Cessation Among Women in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pontifícia Universidade Católica do Paraná (Other); Universidade Estadual de Londrina (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-120606001
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco cessation; women; capacity building
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: The control arm consisted of a home visit by the Community Health Worker scheduling an appointment for the participant to attend the tobacco cessation program at the local Basic Health Unit. The intervention arm consisted of 12-home visits by the Community Health Worker
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention arm consisted of 12-home visits by the Community Health Worker + referring to an appointment for the participant to attend the tobacco cessation program at the local Basic Health Unit.
  Interventions: Behavioral: 12-home visits by the Community Health Worker + referring to an appointment for the participant to attend the tobacco cessation program
- Control (Active Comparator): The control arm consisted of a home visit by the Community Health Worker scheduling an appointment for the participant to attend the tobacco cessation program at the local Basic Health Unit.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Schedule an appointment to attend tobacco cessation at Basic Health Unit
  Arms: Control
Behavioral: 12-home visits by the Community Health Worker + referring to an appointment for the participant to attend the tobacco cessation program — 12-home visits by the Community Health Worker + referring to an appointment for the participant to attend the tobacco cessation program
  Arms: Intervention

SUMMARY:
The overall goal of this renewal is three-fold: (1) to continue to sustain and strengthen the network; (2) to conduct a group randomized controlled trial to assess the efficacy of a theory-based, culturally- and gender-relevant Community Health Worker intervention for Brazilian women "light smokers" that will augment the smoking cessation programs offered through the public health system; and (3) to expand our current Career Development and Research Training Program to the other two major tobacco growing states in order to develop a cadre of well-trained researchers who will continue to develop and implement gender-relevant comprehensive tobacco control strategies at all levels.

DETAILED DESCRIPTION:
An understanding of women and their tobacco-related issues, as well as the need for the development of gender-relevant tobacco control efforts, have been highlighted as priorities in landmark guiding documents published in the past few years (e.g., WHO Framework Convention on Tobacco Control-WHO FCTC). Brazil is the second largest producer of tobacco in the world, and 95% of the tobacco is produced in the three Southern states (Paraná, Santa Catarina, and Rio Grande do Sul). Although, historically, tobacco use among women in developing countries, particularly Latin America, has been relatively low as compared to men, the smoking epidemic is rapidly spreading to women in developing countries, and these three Southern states have the highest prevalence of women smokers in the country. We have established a Network for Tobacco Control among Women in Paraná, Brazil with the purpose of establishing community and institutional capacity to promote gender-relevant tobacco control efforts among women through Community-Based Participatory Research (CBPR) and training. The goals of the network are to reduce tobacco use and exposure to environmental tobacco smoke (ETS) among women in Paraná, and to develop a cadre of well-trained researchers who will continue to address comprehensive tobacco control strategies at multiple levels. The network conducted an epidemiological survey on the prevalence and factors associated with tobacco use among women across the State of Paraná. Based on the results, the network identified four priorities: (1) to implement policy changes to decrease ETS; (2) to understand the health/social issues of women in tobacco farming; (3) to develop and evaluate a comprehensive, culturally- and gender relevant, school-based smoking prevention program; and (4) to improve access and delivery of smoking cessation programs through the public health system with a particular focus on "light smokers" as 74.8% of women smokers in our study reported smoking 10 or less cigarettes/day. The network is currently addressing the first three priorities, including support for legislation, which resulted in Paraná having the strongest indoor tobacco ban in the country.

The overall goal of this renewal is three-fold: (1) to continue to sustain and strengthen the network; (2) to conduct a group randomized controlled trial to assess the efficacy of a theory-based, culturally- and gender-relevant Community Health Worker intervention for Brazilian women "light smokers" that will augment the smoking cessation programs offered through the public health system; and (3) to expand our current Career Development and Research Training Program to the other two major tobacco growing states in order to develop a cadre of well-trained researchers who will continue to develop and implement gender-relevant comprehensive tobacco control strategies at all levels.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Current tobacco user
* 18 years of age
* Living in the randomized neighborhood

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial was gender-relevant to include women only
Enrollment: 338 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Tobacco Cessation | 7 months follow-up
  Our outcome at follow-up, smoking status, was obtained from responses to the question, "Do you smoke any tobacco product?" Respondents could indicate they smoked daily, less than daily, or that they did not smoke. Those who indicated they smoked daily or less than daily were labeled as 'smokers' while those who indicated they did not smoke were labeled 'non-smokers' confirmed by exhaled carbon monoxide level

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data may be shared in the future

REFERENCES:
- [Derived] Scarinci IC, Kienen N, Wiltenburg TD, Bittencourt L, Person SD. Efficacy of a Gender-Relevant Smoking Cessation Intervention Among Women in Brazil: Findings from a Group Randomized Controlled Trial. J Womens Health (Larchmt). 2022 Nov;31(11):1620-1629. doi: 10.1089/jwh.2021.0443. Epub 2022 May 17. PMID 35580140